CLINICAL TRIAL: NCT03449225
Title: Development of a Computer-Aided Genetics Education Module (CAGEM) on Screening and Testing for Fetal Chromosome Conditions and Carrier Status: A Clinical Trial
Brief Title: Prenatal Computer-Aided Genetics Education Module
Acronym: CAGEM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Manesha Putra, MD, Obstetrics and Gynecology Resident Physician, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 115217B3E
Record Dates: First submitted 2018-02-20; First posted 2018-02-28 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Autosomal Recessive Disorder; Aneuploidy
MeSH Terms: conditions — Aneuploidy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): The participant will be given a digital device (IPad or Kindle Fire) to complete a pre-education survey (web-based pre-intervention survey housed on the Qualtrics platform). Once the survey is complete, the participant will proceed with standard education, provided by a resident/physician in the clinic, about prenatal screening and testing for chromosome conditions and for carrier status. Once the standard education has been completed, the participant will be approached to complete a post-education survey which includes questions about knowledge, intent to have or decline screening or testing, and demographic variables.
- Test Arm (Experimental): • The participant she will be given a digital device on which to access the computer aided genetics educational module. Prior to accessing the module, the patient will be asked to complete a pre-education survey (web-based pre-intervention survey housed on the Qualtrics platform). Once she has completed the survey, she will interact with the Computer-Aided Genetic Education Module which is tailored for her clinical situation. Once the participant has completed reviewing the module, she will be asked to complete the web-based post-module survey which includes questions about knowledge, intent to have or decline screening or testing, acceptability of the module, and demographic variables.
  Interventions: Other: Computer-Aided Genetic Education Module

INTERVENTIONS:
Other: Computer-Aided Genetic Education Module — Subjects will be provided with an electronic device to view Computer-Aided Genetic Education Module (CAGEM) software. This is an interactive software designed to provide subjects with tailored information regarding prenatal screening options for carrier status and aneuploidy.
  Arms: Test Arm

SUMMARY:
A standard part of obstetrical care is offering prenatal genetic screening. Numerous professional guidelines have emphasized the importance of pretest counseling for prenatal genetic screenings. Informed consent includes the optional nature of the test, information on the conditions being screened, possible test results, implication of each result, and the type of test offered (screening or diagnostic). This responsibility falls on the physician in a busy clinic. Technology may be able to address this limitation and give consistent pretest counseling for patients waiting for their appointment. This study is looking to evaluate the use of computer-aided genetics education module for facilitating decision making about prenatal genetic screening and testing for fetal chromosome conditions and carrier status.

DETAILED DESCRIPTION:
Rationale Cytogenetic abnormalities are present in nearly 1% of live births, in approximately 2% of pregnancies in women older than 35 years who undergo prenatal diagnosis, and in fully half of all spontaneous, first-trimester abortions. Genetic counseling and screening for cytogenetic abnormalities are an integral part of routine obstetrical care. There are various screening options and strategy available commercially, including screening for the fetus and parental carrier screening. Currently American College of Obstetrics and Gynecology (ACOG) recommends that all pregnant women should be offered screening for fetal aneuploidy. ACOG also recommends panethnic screening for cystic fibrosis, hemoglobinopathies and spinal muscular atrophy carrier status. For other conditions, glycogen storage diseases and fragile X syndrome, the recommendation currently is to screen based on ethnicity and family history. Without thorough counseling, pregnant women may accept multiple screenings without considering the downstream consequences, including anxiety created by additional, sometimes uncertain, information.

Numerous professional societies guidelines have emphasized the importance of pre-test counseling in this setting due to the delicate and complicated nature of genetic conditions. Along with these guidelines, typically minimal recommended information to be provided during a pre-test counseling was included. Generally it involves, the optional nature of the test, general information about condition tested, nature of testing (screening, carrier screening or diagnostic), testing options, possible testing result, implication of each result, cost and availability of genetic counseling should needed. The responsibility of offering these tests and to perform pre-test counseling lie primarily on the obstetrical care providers and has become more burdensome as the number of testing options expands and also due to limited time for discussion during a prenatal care.

Technology may be able to address these limitations. Various studies have evaluated the use of Computerized Decision Aids (CDAs) in facilitating high-quality decision making in various health related contexts with promising results (17-20). CDAs are generally superior to traditional decision aids such as, paper-based or video-based, due to the possibility to tailor CDAs based on the information provided, the ease of information dissemination and also their interactive features which reinforce participation. This study is looking to evaluate the use of computer-based pre-test education for prenatal cytogenetic abnormalities screening.

Statement of Problem Per professional society guidelines, all women should be offered prenatal screening and/or diagnostic testing for fetal aneuploidy (chromosome conditions such as Down syndrome, trisomy 18, trisomy 13, and sex chromosome abnormalities) during pregnancy. Women should also be offered population-based carrier screening but have the option of expanded carrier screening as well. There are an increasing number of testing and screening options available during pregnancy. The obstetrics provider is primarily responsible for ensuring patients are informed about their options and the benefits, risks, and limits of each. These discussions can be time intensive in a setting where the time available is often limited. As such, there is a need to find alternate ways to educate women about their prenatal testing and screening options.

Objectives The overarching purpose of the full project is to determine whether a computer aided genetics education module can improve pregnant women's knowledge about their options for fetal aneuploidy (chromosome) screening and testing and carrier screening and facilitate informed decision making.

The specific aims of the current study are to:

* To develop a computer-aided genetics education module for prenatal cytogenetic abnormalities screening and testing and carrier screening
* To determine the acceptability of the computer-aided genetics educational module for women presenting for care in an obstetrics clinic
* To determine the feasibility of using the computer-aided genetics educational module in a busy obstetrics clinic
* To assess whether use of the module increases knowledge and enhances informed decision making
* To compare the effectiveness of the computer-aided education module to standard care in terms of knowledge gained and impact on decision making

This study will be done in two phases. Phase 1 will involve evaluating the acceptability of the computer-aided genetics education module. Changes will be made to the module based on the feedback obtained. The revised module will then be used for Phase 2. Phase 2 will involve comparing the effectiveness of the computer-aided genetics education module to standard care.

Methodology

A clinician who has access to the daily clinic patient list will identify patients eligible to participate in the study and notify an onsite study team member. Eligible study participants will then be approached by one of the study team members (either a genetic counselor, a genetic counseling student, a medical student, or a maternal-fetal medicine fellow) and be invited to participate in the study. The potential participant will be given the study information sheet and the study team member will review it with her. If the approached participant agrees to take part, participant will be randomized into one of the two arms of the study-control versus tests arm. Randomization will be performed using Qualtrics platform.

* Control arm: The participant will be given a digital device (IPad or Kindle Fire) to complete a pre-education survey (web-based pre-intervention survey housed on the Qualtrics platform). Once the survey is complete, the participant will proceed with standard education, provided by a resident/physician in the clinic, about prenatal screening and testing for chromosome conditions and for carrier status. Once the standard education has been completed, the participant will be approached to complete a post-education survey which includes questions about knowledge, intent to have or decline screening or testing, and demographic variables. Once the post-education survey is completed, the participant will be given a $5 gift card for her time. Participation in the study is then complete.
* Test arm: The participant she will be given a digital device on which to access the computer-aided genetics educational module. Prior to accessing the module, the participant will be asked to complete a pre-education survey (web-based pre-intervention survey housed on the Qualtrics platform). Once she has completed the survey, she will interact with the module which is tailored for her clinical situation. Once the participant has completed reviewing the module, she will be asked to complete the web-based post-module survey which includes questions about knowledge, intent to have or decline screening or testing, acceptability of the module, and demographic variables.
* All responses (control and test) will be recorded using a unique participant identification number in order to pair pre- and post-intervention responses. The identifier will not be linked to any identifiable information. Of note, all subjects will receive standard provider counseling after completion of the study module (standard of care).

Phase 1: During Phase 1, The investigators will assess the acceptability of the computer-aided genetics educational module in our target study population. During this initial phase, The investigators will only be doing the test arm of the study. Quantitative and qualitative responses from the pre- and post-surveys will be obtained from batches of 10 samples; the module will then be optimized based on the qualitative feedback and overall results on the knowledge, acceptability, and informed consent questions. This will be repeated until user acceptability reaches 80% of the maximum score.

The computerized educational module has been developed based on counseling points recommended by the American College of Obstetrics and Gynecology and is based on a previous study investigating computer-aided education. The application can be accessed at https://interva-online.mobi/CAGEM/participant/guestLogin.do?packageId=178

Survey Instruments There are three separate survey instruments, all of which have been developed on the Qualtrics survey platform. The pre-education survey instrument is the same for control and test participants and includes basic knowledge questions about genetic testing and screening for chromosome conditions and carrier status. The questions are based on the standard information that should be presented when providing genetic counseling on these topics.

There are two versions of the post-intervention survey. Both versions include knowledge questions (same as pre-test questions) and demographic questions. The surveys differ in that the survey for those taking part in the test arm include questions about the acceptability of the computer-aided genetics educational module.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant with gestational age of less than 24 weeks
* Good understanding of spoken English

Exclusion Criteria:

* Known history of genetic disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge of Genetics | Participant will be assessed from the time of randomization and again after clinical encounter (and intervention, for the study arm). The total estimated time will be approximately 1 hour since randomization.
  Survey will be used to assess subjects' knowledge on prenatal genetics

SECONDARY OUTCOMES:
Testing Intention | Participant will be assessed from the time of randomization and again after clinical encounter (and intervention, for the study arm). The total estimated time will be approximately 1 hour since randomization.
  Survey will be used to assess subjects' intention to accept or decline

OTHER OUTCOMES:
Software Acceptability | Participant will be assessed from the time after the completion of intervention material usage. This is a one time survey, total estimated time is approximately 10 minutes.
  Survey will be used to assess the software acceptability among subjects

CONTACTS AND LOCATIONS:
Overall Officials: Manesha Putra, MD, Principal Investigator — Wayne State University
Locations (1):
- Hutzel Women's Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided